CLINICAL TRIAL: NCT02637986
Title: The Efficacy of Orally Administrated Probiotic Formula in Preventing a Recurrence of a Urinary Tract Infection During Pregnancy - a Prospective Randomized Double Blind Placebo-control Study
Brief Title: The Efficacy of Orally Administrated Probiotic Formula in Preventing a Recurrence of a Urinary Tract Infection During Pregnancy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigatore decided not to proceed with this study
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0173-13-EMC
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Urinary Tract Infections (UTIs)
MeSH Terms: conditions — Urinary Tract Infections | interventions — methenamine hippurate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ARM A - suffered from one episode of UTI (Experimental): Women who suffered from one episode of UTI during pregnancy before recruitment
  Interventions: Dietary Supplement: Urex Plus - containing L. rhamnosus GR-1 and L. reuteri RC-14
- ARM A - suffered from one episode of UTI - placebo (Placebo Comparator): Women who suffered from one episode of UTI during pregnancy before recruitment
  Interventions: Other: Placebo - capsule with no active ingredient
- ARM B -suffered from more than one episode of UTI (Experimental): women who suffered from more than one episode of UTI or one episode of pyelonephritis during pregnancy before recruitment
  Interventions: Dietary Supplement: Urex Plus - containing L. rhamnosus GR-1 and L. reuteri RC-14
- ARM B -suffered from more than one episode of UTI - placebo (Placebo Comparator): women who suffered from more than one episode of UTI or one episode of pyelonephritis during pregnancy before recruitment
  Interventions: Other: Placebo - capsule with no active ingredient

INTERVENTIONS:
Dietary Supplement: Urex Plus - containing L. rhamnosus GR-1 and L. reuteri RC-14 — 2 capsules will be given per day
  Arms: ARM A - suffered from one episode of UTI; ARM B -suffered from more than one episode of UTI
Other: Placebo - capsule with no active ingredient — 2 capsules will be given per day
  Arms: ARM A - suffered from one episode of UTI - placebo; ARM B -suffered from more than one episode of UTI - placebo

SUMMARY:
Background: Urinary tract infections (UTIs), the most common infection in pregnancy,are associated with several maternal and fetal complications, including maternal septic shock, preterm labor, intrauterine growth restriction and intrauterine fetal death. Thus, the prevention of UTIs in pregnancy is a very important goal. Several studies have suggested that alterations in the vaginal flora were associated with recurrent UTIs, and probiotic administrations may have a role in preventing those infections. Nevertheless, this has never been tested in pregnant women.

DETAILED DESCRIPTION:
Background: Urinary tract infections (UTIs), the most common infection in pregnancy,are associated with several maternal and fetal complications, including maternal septic shock, preterm labor, intrauterine growth restriction and intrauterine fetal death. Thus, the prevention of UTIs in pregnancy is a very important goal. Several studies have suggested that alterations in the vaginal flora were associated with recurrent UTIs, and probiotic administrations may have a role in preventing those infections. Nevertheless, this has never been tested in pregnant women.

Working hypothesis and aims:Administration of oral probiotic formula to pregnant women,which suffered from at least one episode of UTI, will reduce the recurrence of future UTIs events.

Methods: A prospective randomized double blind placebo-control study. Pregnant women which suffered from at least one event of UTI during pregnancy will be divided into 2 research arms:

ARM A - women who suffered from one episode of UTI during pregnancy before recruitment: after antibiotic treatment achieving a sterile bacterial urine culture, these patients will be divided into a research group which will receive the probiotic formula Urex Plus containing L. rhamnosus GR-1 and L. reuteri RC-14, and a control group, which will receive a placebo, twice a day until delivery.

ARM B - women who suffered from more than one episode of UTI or one episode of pyelonephritis during pregnancy before recruitment will receive a preventive antibiotic treatment until delivery. Similarly to ARM A, after achieving a sterile bacterial urine culture, those women, will be divided into a research group, which will receive the probiotic formula Urex Plus, and a control group, which will receive a placebo twice a day until delivery.

Once a month and with symptoms, urine culture will be taken in all of the study arms. Vaginal swab test will also be taken to detect the presence of abnormal vaginal flora and semi-quantitative assessment of vaginal lactobacilli.

Data regarding the rate of recurrent UTIs, time until infection, average number of infections, the rate of pyelonephritis infections and obstetrical and neonatal outcomes will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* Pregnant women who suffered from at least one episode of UTI
* Women less than 34th week of gestation at the time of the enrollment
* Urine culture is sterile in the beginning of the study

Exclusion Criteria:

* Immunocompromised women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
The rate of women who developed UTI after receiving probiotic formula versus placebo. | 1 year
  The rate of women who developed UTI after receiving probiotic formula versus placebo.

SECONDARY OUTCOMES:
Duration of time from the beginning of study until an episode of UTI. | 1 year
The number of UTIs during pregnancy. | 1 year
The rate of women who suffer from bacteruria, cystitis and pyelonephritis. | 1 year
The rate of women who suffer from obstetrical outcomes (preterm labor, intrauterine growth restriction). | 1 year
Adverse effects of the probiotic capsules versus placebo | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Enav Yefet, MD/PhD, Principal Investigator — Emek Medical Center

IPD SHARING:
Plan to Share IPD: No